CLINICAL TRIAL: NCT01946763
Title: Does Pre-operative Patients' Education Facilitates Emergence of Anesthesia Following Bariatric Surgery?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Procare Riaya Hospital (Other)
Responsible Party: Principal Investigator, Ahed ZEIDAN, Anesthesiologist, Procare Riaya Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRH06
Record Dates: First submitted 2013-06-03; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- safety of Anesthesia (No Intervention): No pre operative education
- Behavioral : pre operative education (Experimental): Behavioral pre operative education
  Interventions: Behavioral: pre operative education

INTERVENTIONS:
Behavioral: pre operative education — Patients will be randomized in 2 groups (G1: educated, G2:non-educated) In the operating room and before starting anesthesia G1 will receive a pre operative education about anesthesia emergence, recovery and extubation.
  Arms: Behavioral : pre operative education
Behavioral: pre operative education
  Arms: Behavioral : pre operative education

SUMMARY:
The recovery and emergences from anesthesia is a critical phase. Previous studies focused on pharmological and anesthetics techniques to improve the quality of this stage (duration, complications).

In this study, our first aim is to test the impact of pre operative education on the post operative recovery for morbidly obese patient underwent laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
The purpose of our study is to compare post operative immediate recovery and emergence for educated and non educated morbidly obese patients underwent laparoscopic bariatric surgery.

Elligibles patients are informed and consented by anesthesiologist. Patients are randomized in 2 groups (G1: educated, G2:non-educated) Patient of G1 are educated in OR before starting anesthesia. This education includes : information about anesthesia emergence, recovery and extubation.

Anesthesia and education are conducted by the same anesthesiologist. All patients are operated by the same surgeon. All patients receive same balanced general anesthesia protocol. The recovery starts immediately after the end of the procedure, when the patient has BIS ≥90 and TOF≥9.

Recovery assessment and data recording is done by a blinded anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 18 years old.
* ASA 2.
* BMI more than 35.
* scheduled for laparoscopic sleeve gastrectomy or gastric bypass surgery.

Exclusion Criteria:

* Renal impairment.
* Hepatic dysfunction.
* Alcohol or drug abuse.
* Disabling Central nervous or cerebrovascular diseases.
* Treatment with opioids or any psychoactive medication.
* Inappropriate Mini mental state exam.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Quality of anesthesia recovery | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahed Zeidane, MD, Principal Investigator — Procare Riaya Hospital
Locations (1):
- Procare Riaya Hospital, Khobar, Eastern Province, Saudi Arabia